CLINICAL TRIAL: NCT05738239
Title: Application of Photo-biomodulation as Part of Multimodal Analgesia to Improve Pain Relief and Wound Healing for Patients Having Elective Caesarean Section: a Randomized Controlled Trial
Brief Title: Photo-biomodulation Therapy for Pain Relief After Caesarean Section
Acronym: PBMT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PBMT-2023
Record Dates: First submitted 2023-01-27; First posted 2023-02-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Pain
Keywords: Postoperative wound pain; Caesarean section; Photo-biomodulation therapy; Low-level LASER; Chronic post-surgical pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: Active PBMT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Application of photo-biomodulation
  Interventions: Device: Laser therapy
- Placebo (Placebo Comparator): Inactive PBMT
  Interventions: Device: Laser therapy

INTERVENTIONS:
Device: Laser therapy — Biological effects of low-level LASER therapy have been studied for various clinical indications, including musculoskeletal conditions and some acute pain conditions. PBMT includes low level LASER (works on pain) and light-emitting diodes (LED) (works on wound healing).

SUMMARY:
C-sections may result in a lot of pain that is distressing to the mother, and can impact bonding with the baby. Although there are medications used to treat strong pain, they are not good to use after C-sections because they can affect the baby. There is a need for a pain management option that can reduce the use of medications. The investigators are testing the effects of a combined light and laser device (photo-biomodulation therapy; PBMT), used on the wound twice daily, with respect to pain right after surgery, and pain that lasts longer than 6 weeks after surgery.

DETAILED DESCRIPTION:
Background Caesarean section (CS) is the most common inpatient surgical procedure performed in Canada, with an average duration of stay of 2.7 days. Its rate continues to increase; from 28.2% in 2016-2017 to 31.0% in 2020-2021. CS is commonly performed under neuraxial anesthesia (spinal or epidural) with majority of elective CSs being carried out under spinal anesthesia. It is associated with moderate to severe pain in most women and is more severe within the first 2 days. In a large cohort study involving 1288 parturients including 391 women having caesarean delivery, the mean pain score (standard deviation) was 4.7 (2.0). In another prospective study of 195 women having elective CS under spinal anesthesia, the median (interquartile range) visual analogue score (0-100 scale) with movement was 53 (32-72). Avoidance of pain during and after CS was noted to be the topmost priority among women. Significant pain after CS not only causes maternal distress but interferes with neonatal bonding and furthermore predisposes a woman for persistent pain and postpartum depression.

Chronic or persistent pain after CS can be an important problem. As per the International Association for the Study of Pain (IASP), chronic post-surgical pain (CPSP) is defined as pain that develops on increases after a surgical procedure as identified at three months or more after surgery; localized to the area of surgery or projected to the innervation territory; and pain that is not explained by an infection, malignancy, a pre-existing pain condition or any other alternative cause.

A prospective study of 527 women noted an incidence of 18.3 %, 11.3 % and 6.8 %, respectively at 3, 6 and 12 months, and observed that more severe pain during movement within 24 h of surgery and preoperative depression were predictive of pain persistence at 6 months. A more recent prospective study of 462 women (among 621) notes an incidence of 25.5% (95% CI: 21.8-29.7) at 90 days. Presurgical anxiety (adjusted relative risk [RR] 1.03; 95%CI: 1.01-1.05), smoking (adjusted RR 2.22; 95%CI: 1.27-3.88) and severe pain in the early postoperative period (adjusted RR 2.79; 95%CI: 1.29-6.00) were predictive of CPSP. Overall, the incidence of CPSP after CS can vary between 4% to 41.8% and generally decreases over time. Although factors associated with its development are noted to be inconsistent in studies, presence of severe pain in the first 1-2 days after surgery can be noted as the most commonly identified factor. CPSP can lead to significant maternal distress, suffering, continued need and potential long-term exposure to opioids, and post-partum depression (PPD). PPD is one of the commonest maternal long-term complication after childbirth, with an incidence of around 13%, as noted in published studies and also in a large observational study. History of preoperative depression and post-surgical pain can influence the incidence of PPD. In a longitudinal study of 1288 women, there was a threefold increase in the odds of PPD (at 8 weeks) in women having severe acute postpartum pain. In studies, screening for PPD is commonly performed using the Edinburgh Postnatal Depression Scale consisting of 10 questions, and a threshold of >12 is considered as positive for PPD.

Photo-biomodulation therapy (PBMT) and pain relief Biological effects of low-level LASER therapy have been studied for various clinical indications. Over the years the differential effects of light emitting diodes (LEDs) in causing stimulatory effects including wound healing, epithelialization and angiogenesis, and deeper inhibitory doses of radiation by LASER in modulating pain signals have been recognized (19). As per the American Society for Laser Medicine and Surgery the term photo-biomodulation should be used, and PBMT is defined as a "form of light therapy that utilizes non-ionizing forms of light sources including LASERS, LEDs, and broadband light, in the visible and near infrared spectrum". PBMT has been used in many musculoskeletal conditions and in some acute pain conditions. Its proposed mechanism of action on pain and wound healing includes increased production of anti-inflammatory cytokines and local neo-angiogenesis apart from other actions.

Considering the existing limitations in multimodal analgesia and a concerted need to avoid opioids in this context, there is a greater need for non-pharmacological strategies. Photo-biomodulation therapy (PBMT) can improve pain control and wound healing. By using PBMT after surgery, the investigators have the potential to achieve better pain control and postoperative outcomes. The study aims to evaluate the effectiveness of PBMT as part of existing multimodal analgesia, so that it can be demonstrated as appropriate for clinical use. This will result in improved maternal satisfaction and wound healing; decrease the use of perioperative opioids; potentially influence a decrease in the incidence of postpartum depression and persistent pain; and overall lead to better postoperative outcomes thereby decreasing healthcare costs.

Objectives Primary objective: To evaluate the effect of PBMT as part of a multimodal analgesia on post-surgical pain burden using pain scores with movement, after elective caesarean deliveries. Secondary objectives: To evaluate the effect of PBMT on the following outcomes during the hospital stay (up to 48 hours) after surgery: 1) Pain scores at rest; 2) The percentage of patients with moderate and severe pain; 3) The dose of total opioid used in mg of oral morphine equivalents; 4) The incidence of opioid-related adverse including nausea-vomiting and sedation, and 5) Patient satisfaction at hospital discharge. To evaluate the effect of PBMT on the following outcomes at 6 weeks after surgery: 6) The incidence of surgical wound infection and delayed wound healing; 7) The incidence of persistent pain around the surgical site, 8) The incidence and severity of PPD, and lastly 9) Any adverse effects related to the use of PBMT at any time during the study. Tertiary objectives: In all patients, to evaluate the following outcomes at 3 months after surgery: 1) incidence of chronic post-surgical pain, and 2) incidence of delayed wound healing or wound infection at 3 months after surgery, 3) incidence of PPD, and lastly 4) Any adverse effects related to the use of home based PBMT.

Design Placebo-controlled two-arm parallel-design randomized controlled trial Screening and Baseline data collection At each site there are typically 2-3 women booked for elective CS each day, with approximately 8-10 surgeries per week. Patients will be approached on the morning of surgery and informed about the study. Patients willing to participate will be consented along with collection of baseline study variables.

Study interventions Study Group Patients will have 5 treatment sessions of PBMT provided by a trained research nurse; 4 hrs after the CS, then morning (8 am), and evening (7 pm) of postoperative day (POD) 1 and 2. Each session will involve LED therapy (7 minutes) using DUO 240 LED (red at 660 nm and near infrared at 840 nm) applied parallel to the abdominal incision scar, followed by simultaneous spot treatment using the BIOFLEX LDR-100 laser probe (660 nm red light) and the LD1-200 laser probe (825 nm near infrared light), applied at the incision wound edges, for a total treatment time of 10 minutes.

Placebo Group Patients will have 5 treatment sessions following the same schedule as above, with non-effective doses of LED array and LASER therapy.

Data Collection and Follow-Up All patients will be followed by a blinded research assistant for 7 time points during their hospital stay and relevant outcomes will be collected; evening of surgery (8-9 pm); on POD 1 and 2 at morning (9-10 am), noon (12-1 pm), and evening (8-9 pm). All patients will also be contacted at 6 weeks in person, to coincide with their expected follow-up visit with their physician and relevant outcomes will be collected.

At the 6-week follow-up, patients with either persisting pain or delayed wound healing will be provided with the option of using home-based PBMT as per the randomized groups (active or placebo), 3-5 times/day until 3 months after surgery.

Sample size considerations Sample size was estimated based on a mixed model of repeated measures with general correlation structure (30). A mean score of 4.7 and SD of 2 was considered for the control group (3) and a mean difference of 1 point or more in 0-10 NRS was considered as the treatment effect. Using an alpha of 0.05 and power of 90%, and an attrition of 5%, our sample size would be 90 per group.

Data analysis According to the intention-to-treat principle and reported as per the CONSORT guidelines. Primary outcome of pain intensity for repeated measures will be analyzed using a generalized estimating equations model (GEE), with pain scores modeled as a function of time, with the use of appropriate model and correlation structure. Secondary and tertiary outcomes will be analyzed with appropriate logistic and linear regression models after adjusting for baseline variables that are known to influence these outcomes. For all, statistical significance will be considered using a 2-sided test with p-value is <0.05. All analyses will be performed in R version 4.2.1. The investigators will perform a subgroup analysis for outcomes collected at 3 months based on the patients who used home based PBMT.

Ethical considerations This trial will be conducted in compliance with the protocol, principles laid down in the Declaration of Helsinki, Good Clinical Practice (GCP), as defined by the International Conference on Harmonisation (ICH). This protocol will be reviewed and approved by the Hamilton Integrated Research Ethics Board (HiREB) prior to commencement of the trial.

ELIGIBILITY:
Inclusion Criteria:

• Women aged ≥18 years with planned C-Section under spinal anesthesia.

Exclusion Criteria:

* Not willing
* Language barrier or cannot communicate in English.
* History of chronic ongoing pain needing daily opioid medications
* High risk or twin/multiple pregnancy
* C-Section planned under a general anesthetic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Evening of surgery (8-9 pm)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 1, morning (9-10 am)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 1, noon (12-1 pm)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 1, evening (8-9 pm)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 2, morning (9-10 am)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 2, noon (12-1 pm)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
Pain intensity with movement (elicited by asking the patient to move from supine to sitting position) using 0-10 Numerical Rating Scale | Postoperative day 2, evening (8-9 pm)
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.

SECONDARY OUTCOMES:
Pain scores at rest | 7 time points: evening of surgery (8-9 pm); POD 1 and 2 at morning (9-10 am), noon (12-1 pm), and evening (8-9 pm).
  The 0-10 Numerical Rating Scale (NRS) (0=no pain, 10=worst possible pain, patient reported.
The percentage of patients with moderate and severe pain | Average of pain scores from 7 time points: evening of surgery (8-9 pm); POD 1 and 2 at morning (9-10 am), noon (12-1 pm), and evening (8-9 pm).
  Patients with average resting pain score of >4/10 on the Numerical Rating Scale during their hospital stay
Total opioid dose used in hospital | 3 days: Day of surgery until discharge from hospital
  All opioids used will be converted into oral morphine milligram equivalents for comparison
Incidence of patients with clinically important postoperative nausea/vomiting (PONV). | 3 days: Day of surgery until discharge from hospital at 7 time points: evening of surgery (8-9 pm); POD 1 and 2 at morning (9-10 am), noon (12-1 pm), and evening (8-9 pm).
  Clinically important postoperative nausea/vomiting (PONV) measured using a validated PONV intensity scale,
  Wengritzky R, Mettho T, Myles PS, Burke J, Kakos A. Development and validation of a postoperative nausea and vomiting intensity scale. Br J Anaesth. 2010;104(2):158-66
Incidence of severe sedation | 3 days: Day of surgery until discharge from hospital at 7 time points: evening of surgery (8-9 pm); POD 1 and 2 at morning (9-10 am), noon (12-1 pm), and evening (8-9 pm).
  Patients with grade 3 and above in the Pasero Opioid-induced Sedation scale (grade 3= frequently drowsy, arousable but drifts off to sleep during conversation)
  Nisbet AT, Mooney-Cotter F. Comparison of selected sedation scales for reporting opioid-induced sedation assessment. Pain Manag Nurs. 2009;10(3):154-64
Patient satisfaction at hospital discharge | Postoperative day 3
  Measured using a 0-10 scale (0=least satisfied; 10=most satisfied), patient reported
Wound healing | 6 weeks postoperatively
  Number of patients with physician identified i) delayed healing and ii) surgical skin site infection (as per the CDC criteria)
  Network NHS 2023;Pages. Accessed at Centers for Disease Control and Prevention at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf on January 19 2023.
Incidence of persistent pain | 6 weeks postoperatively
  Elicited as Yes/No and intensity recorded using 0-10 NRS. (0=no pain, 10=worst possible pain)
Incidence of postpartum depression | 6 weeks postoperatively
  Considered as positive if the Edinburgh Postnatal Depression Scale (EPDS) score is ≥12 The 10-question Edinburgh Postnatal Depression Scale (EPDS) helps identify patients at risk for "perinatal" depression. Scores range from 0 (not at all at risk) to 30 (highest possible risk). Scores of 12 and over are considered as postpartum depression
Incidence of adverse effects due to PBMT | Any time point in the study (POD0 to 3-month follow-up)
  Incidence of any skin allergy or injury or reaction to PBMT treatment

OTHER OUTCOMES:
Incidence of chronic postsurgical pain | 3 months postoperatively
  As per International Association for the Study of Pain (IASP) definition:
  Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019;160(1):45-52
Incidence of delayed or abnormal wound healing or surgical site infection | 3 months
  Patients will be asked about any ongoing issue and evaluated with a physician follow up if appropriate. Number of patients with physician identified i) delayed healing and ii) surgical skin site infection (as per the CDC criteria) :
  Network NHS 2023;Pages. Accessed at Centers for Disease Control and Prevention at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf on January 19 2023
Incidence of postpartum depression | 3 months
  Considered as positive if the Edinburgh Postnatal Depression Scale (EPDS) score is ≥12
Incidence of any adverse effects related to the use of home-based PBMT | 3 months
  including incidence of any skin allergy or injury or reaction to PBMT treatment

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Shanthanna, MD, Principal Investigator — SJHH and McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisenach JC, Pan PH, Smiley R, Lavand'homme P, Landau R, Houle TT. Severity of acute pain after childbirth, but not type of delivery, predicts persistent pain and postpartum depression. Pain. 2008 Nov 15;140(1):87-94. doi: 10.1016/j.pain.2008.07.011. Epub 2008 Sep 24. PMID 18818022
- [Result] Cheng K, Martin LF, Slepian MJ, Patwardhan AM, Ibrahim MM. Mechanisms and Pathways of Pain Photobiomodulation: A Narrative Review. J Pain. 2021 Jul;22(7):763-777. doi: 10.1016/j.jpain.2021.02.005. Epub 2021 Feb 23. PMID 33636371